CLINICAL TRIAL: NCT05066165
Title: Phase 1/2a, Single Dose Study Investigating NTLA-5001 in Subjects With Acute Myeloid Leukemia
Brief Title: Study Investigating NTLA-5001 in Subjects With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Pivoting to an allogeneic version of this program currently in preclinical development.
Sponsor: Intellia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ITL-5001-CL-001
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Results first posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: NTLA-5001; cell kinetics; Pharmacodynamics; clustered regularly interspaced short palindromic repeats; CRISPR; AML; Acute Myeloid Leukemia; TCR T Cell Therapy; Autologous; Leukemia; Neoplasms; Immune System Diseases; Immunoproliferative Disorders
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Neoplasms; Immune System Diseases; Immunoproliferative Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: NTLA-5001 (Experimental): Up to three escalation cohorts in phase 1 followed by one expansion cohort in phase 2. Subjects have AML and bone marrow blast count <5%, administered by IV infusion following lymphodepleting chemotherapy.
  Interventions: Genetic: Arm 1: NTLA-5001
- Arm 2: NTLA-5001 (Experimental): Up to three escalation cohorts in phase 1 followed by one expansion cohort in phase 2. Subjects have AML and bone marrow blast count ≥5%, administered by IV infusion following lymphodepleting chemotherapy.
  Interventions: Genetic: Arm 2: NTLA-5001

INTERVENTIONS:
Genetic: Arm 1: NTLA-5001 — Autologous WT1-directed TCR T cells engineered ex vivo using CRISPR/Cas9 as intravenous infusion after pre-conditioning chemotherapy.
  Cyclophosphamide and Fludarabine will be administered on Day -5, -4, and -3 as intravenous infusion.
  Arms: Arm 1: NTLA-5001
Genetic: Arm 2: NTLA-5001 — Autologous WT1-directed TCR T cells engineered ex vivo using CRISPR/Cas9 as intravenous infusion after pre-conditioning chemotherapy.
  Cyclophosphamide and Fludarabine will be administered on Day -5, -4, and -3 as intravenous infusion.
  Arms: Arm 2: NTLA-5001

SUMMARY:
This study will be conducted to evaluate the safety, tolerability, cellular kinetics (CK), activity, and pharmacodynamics (PD) of NTLA-5001 in participants with Acute Myeloid Leukemia (AML).

DETAILED DESCRIPTION:
This 2-part first in human (FIH) study is comprised of two open-label arms. It is a multi-center, Phase 1/2a study evaluating the safety and activity of NTLA-5001 in subjects with persistent or recurrent Acute Myeloid Leukemia after first-line or later therapy.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

* Has AML as defined by World Health Organization
* Has detectable disease following first-line therapy
* Is ≥ 18 years of age.
* Carries the human leukocyte antigen-A0201 (HLA-A*02:01) allele.
* Has ECOG performance status of 0 to 1.
* Has adequate absolute total lymphocyte count
* Has adequate cardiac, renal, and liver organ function

Exclusion Criteria (abbreviated):

* Has received AML-directed therapy or immunomodulatory therapy within a specified window prior to study entry.
* Has received allogeneic hematopoietic cell transplant within 84 days, with ongoing GVHD, with recent DLI, or on active immunosuppression.
* Has CNS involvement by tumor.
* Has severe autoimmunity requiring immunomodulatory therapy.
* Has active disseminated intravascular coagulation (DIC), bleeding or coagulopathy.
* Has leukocytosis ≥ 20,000 blasts/μL despite hydroxyurea or has rapidly progressive disease
* Has human immunodeficiency virus (HIV) infection, or any uncontrolled infection.
* Female subjects are pregnant or breastfeeding; or are of childbearing potential and are unwilling to use protocol specified method of contraception.
* Male subjects who have female partners of childbearing potential and are unwilling to use protocol specified method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - Research Site 2, Los Angeles, California
  - Research Site 5, Tampa, Florida
  - Research Site 1, Boston, Massachusetts
  - Research Site 6, Portland, Oregon
  - Research Site 3, Houston, Texas
  - Research Site 4, Milwaukee, Wisconsin
- United Kingdom (4):
  - Research Site 10, Leeds
  - Research Site 8, London
  - Research Site 9, London
  - Research Site 7, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 participants were enrolled at 3 sites in one country. A total of 2 participants received the product at Dose Level 1 in the Dose Escalation phase. The first participant was enrolled on 17 December 2021 and the last participant was enrolled on 21 July 2022. Dose escalation phase did not proceed beyond Dose Level 1. Dose Expansion phase was not initiated.
Pre-assignment Details: Six participants were enrolled in the study (signed informed consent and underwent leukapheresis), but only two participants were dosed (administered Dose Level 1).
Groups:
- Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow: Arm 1: NTLA-5001: Autologous WT1-directed TCR T cells engineered ex vivo using CRISPR/Cas9 as intravenous infusion after pre-conditioning chemotherapy. The participant was administered Dose Level 1.
- Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow: Arm 2: NTLA-5001: Autologous WT1-directed TCR T cells engineered ex vivo using CRISPR/Cas9 as intravenous infusion after pre-conditioning chemotherapy. The participant was administered Dose Level 1.
Period: C1:DoseLevel1 Assignment
Arm/Group | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow
Started | 1 | 5
Completed | 1 | 1
Not Completed | 0 | 4
Not completed — Pivoting to an allogeneic version of this program | 0 | 4
Period: C1:DoseLevel1 Dosed Participants (W1-16)
Arm/Group | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Death | 1 | 1
Period: Cohort2:Dose Level 2
Arm/Group | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Five participants were enrolled in Arm 2, but only one was dosed.
Groups:
- Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow: Arm 1: NTLA-5001: Autologous WT1-directed TCR T cells engineered ex vivo using CRISPR/Cas9 as intravenous infusion after pre-conditioning chemotherapy.
- Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow: Arm 2: NTLA-5001: Autologous WT1-directed TCR T cells engineered ex vivo using CRISPR/Cas9 as intravenous infusion after pre-conditioning chemotherapy.
- Total: Total of all reporting groups
Arm/Group | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow | Total
Number analyzed (Participants) | 1 | 5 | 6
Age, Continuous [Median (Full Range); unit: years] | 68 [68 to 68] | 57 [41 to 74] | 59 [41 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 5 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 5 | 6
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 37.7 (0) | 24.3 (6.63) | 26.5 (8.07)
Height [Mean (Standard Deviation); unit: cm] | 190.0 (0) | 170.2 (9.18) | 173.5 (11.52)
Weight [Mean (Standard Deviation); unit: kg] | 136.0 (0) | 71.3 (24.79) | 82.1 (34.50)

OUTCOME MEASURES:

1. Primary Outcome: Participants That Experienced Dose-limiting Toxicities (DLTs)
Description: DLTs were defined as events with onset within 28 days of infusion. AEs were collected from time of informed consent through the Week 112 visit. AEs were coded using Medical Dictionary for Regulatory Activities (MedDRA) version 24.0. Severity of AEs was assessed by the investigator using the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 toxicity grading criteria. The measure reported below for the primary outcome consists of DLT data only. Adverse events are reported in the Adverse Event section of this presentation.
Time Frame: Primary DLT assessment from NTLA-5001 infusion up to 28 days post-infusion
Population: The Safety Analysis Set (defined as all participants who received NTLA-5001) was used for this presentation.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

2. Secondary Outcome: Frequency of NTLA-5001 T-cell Receptor (TCR) Transgene Copy Number in the Peripheral Blood
Description: Frequency of edited TCR transgene copy number in the peripheral blood of the participants was determined by droplet digital polymerase chain reaction (ddPCR).
Time Frame: From NTLA-5001 infusion up to 4 weeks post-infusion
Population: The Cell Kinetics Analysis Set (defined as all participants who received NTLA-5001 and have at least one evaluable cell kinetics sample) was used for this presentation.
Measure: Mean (Standard Deviation); unit: copy/ng gDNA
Arm/Group | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow
Number analyzed (Participants) | 1 | 1
copy/ng gDNA | NA (NA) — Transgene in all collected patients' samples were below limit of quantification or negative | NA (NA) — Transgene in all collected patients' samples were below limit of quantification or negative

3. Secondary Outcome: Persistence of NTLA-5001 T Cell Receptor (TCR) Transgene Copy in Peripheral Blood
Description: Persistence of edited TCR transgene copy in the peripheral blood of the participants determined by ddPCR.
Time Frame: From NTLA-5001 infusion up to 4 weeks post-infusion
Population: as for outcome 2
Measure: Number; unit: Days
Arm/Group | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow
Number analyzed (Participants) | 1 | 1
Days | NA — Transgene levels and Persistence were not quantifiable, as no participant had measurable values for edited TCR transgene copies | NA — Transgene levels and Persistence were not quantifiable, as no participant had measurable values for edited TCR transgene copies

4. Secondary Outcome: Tumor Response in Participants With AML
Description: Rate of objective response, where response is complete response without measurable residual disease (CRMRD-) (Arm 1). Rate of objective response, where response is CRMRD-, complete response, complete remission with incomplete hematologic recovery, morphologic leukemia-free state, and partial remission (Arm 2).
Time Frame: From NTLA-5001 infusion up to 4 weeks post-infusion
Population: The Safety Analysis Set (defined as all participants who received NTLA-5001) was used for presentations of disease response data.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

5. Secondary Outcome: Response Duration in Participants With AML
Description: Bone marrow results were planned to be used to determine the duration of response / remission (DOR) for subjects with objective response, from first response until MRD was measured above the lower level of detection for the central laboratory assay, or death from any cause, whichever occurred first (Arm 1). Bone marrow results were planned to be used to determine DOR for subjects with composite CR, from first response to progression or death due to any cause, whichever occurred first (Arm 2).
Time Frame: From NTLA-5001 infusion up to 4 weeks post-infusion
Population: as for outcome 4
Measure: Median (Standard Deviation); unit: Weeks
Arm/Group | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow
Number analyzed (Participants) | 1 | 1
Weeks | NA (NA) — Both participants experienced disease progression at the first assessment | NA (NA) — Both participants experienced disease progression at the first assessment

6. Secondary Outcome: Disease Progression in Participants With AML
Description: Bone marrow results were used to determine the time to clinical progression. Progressive disease was defined as an increase from baseline of at least 25% of bone marrow blasts or an absolute increase of at least 5,000 cells/μL in the number of circulating leukemia cells
Time Frame: From NTLA-5001 infusion up to 4 weeks post-infusion
Population: as for outcome 4
Measure: Median (Standard Deviation); unit: Weeks
Arm/Group | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow
Number analyzed (Participants) | 1 | 1
Weeks | NA (NA) — Both participants experienced disease progression at the first assessment | NA (NA) — Both participants experienced disease progression at the first assessment

ADVERSE EVENTS:
Time Frame: From the date of NTLA-5001 infusion up to 16 weeks post-infusion.
Description: Safety population = all participants who received NTLA-5001.
Arm/Group | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow (N=1) | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: NTLA-5001 Participants With AML Blasts < 5% of Bone Marrow (N=1) | Arm 2: NTLA-5001 Participants With AML Blasts ≥ 5% of Bone Marrow (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Affect lability (Psychiatric disorders) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated by the Sponsor due to a strategic business decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT05066165/Prot_001.pdf
  • Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT05066165/SAP_002.pdf